CLINICAL TRIAL: NCT06055309
Title: Behavioral Pharmacology of Cannabis in Older Adults: A Pilot Study
Brief Title: Behavioral Pharmacology of Cannabis in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 275234
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Health Services for the Aged
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Within-subject design
Masking Description: brownies will contain different doses of cannabis product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabis (up to three doses) (Experimental): Brownies containing a dose of cannabis
  Interventions: Drug: Cannabis (up to three doses)

INTERVENTIONS:
Drug: Cannabis (up to three doses) — a dose of cannabis will be baked into brownies

SUMMARY:
This study examines the effects of cannabis on mood, cognitive and psychomotor performance, balance and vital signs in older adults.

DETAILED DESCRIPTION:
The overarching aims of this pilot study are to determine the dose-related effects of cannabis and explore feasibility and acceptability of conducting a rigorous behavioral pharmacology study in this population. Using a within-subject design in older adults (55-70 years), this study will (1) determine acute dose-related effects of cannabis on physiological, subjective, cognitive, and psychomotor measures and (2) explore acceptability/feasibility of this approach among older adults in order to refine procedures for future studies. Volunteers (55-70 years) will undergo three 7.5-hour experimental sessions conducted one week apart, in which they receive cannabis containing various oral doses of tetrahydrocannabinol (THC) / cannabidiol (CBD) administered in a brownie formulation and the following are assessed: 1) self-reported and/or observer ratings of positive and negative subjective effects; 2) performance effects, measured by reaction time, coordination, and cognitive impairment; and 3) cardiovascular effects. Participants will be contacted the day after each session for feedback on the acceptability of session length, types, number and duration of tasks and any adverse events. Reasons for dropout will also be sought to determine whether study procedures impacted attrition. Findings will: 1) provide investigative team with the hands-on research cannabis research experience; 2) elucidate the optimal THC dose range; and 3) determine the most feasible/acceptable study design in older adults that will inform further rigorous studies examining acute and chronic administration of cannabis formulations among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of marijuana use with no serious adverse effects
* Negative urine toxicology screen for psychoactive drugs (cocaine, fentanyl, methadone, opiates, buprenorphine, methamphetamine, amphetamines, barbiturates, oxycodone, benzodiazepines, phencyclidine, and THC) and CBD
* Negative breath alcohol concentration
* Report ≥1 year abstinence from nicotine and tobacco
* Report ≥1 month of abstinence from THC- and CBD- containing products and be willing to abstain from these products for the study duration
* Blood pressure (BP) reading ≤140/90 and ≥110/70 at the time of screening
* Read and understand English (because assessments are validated in English)
* Menopause as defined as no reported menstruation for ≥12 months (females only)
* Negative urine pregnancy test (females only)
* Stable medical conditions controlled by non-psychoactive medications that do not alter THC/CBD metabolism (e.g., hypertension under control with certain antihypertensives; type II diabetes controlled by metformin)

Exclusion Criteria:

* A history of moderate to severe substance use disorders (SUDs) (except tobacco), according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), and no recent history (≥1 year) of SUD
* Current tobacco/nicotine use
* ECG abnormalities at screening including but not limited to: bradycardia (<55 beats per minute); prolonged QTc interval (>450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block; pre-existing severe gastrointestinal narrowing (pathologic or iatrogenic)
* Have a serious and uncontrolled medical condition (major cardiovascular, renal, endocrine, or hepatic disorder) including a history of serious head trauma or neurological disorder (e.g., seizure disorder)
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for lifetime psychosis, schizophrenia, or bipolar disorder or current major depressive disorder, suicidality (e.g., last month suicidal ideation or suicide attempt in past year, as measured by Columbia Suicide Severity Rating Scale) or have significant psychiatric symptoms of another disorder
* Diagnosis of a cognitive disorder (Alzheimer's Disease, dementia) or a score of <25 on the Montreal Cognitive Assessment (MoCA) for Dementia during screening
* Currently taking any prescribed medication for a psychiatric disorder
* Current use of over-the-counter medication or prescription psychoactive drugs that would be expected to have major interaction with THC (e.g., warfarin, serotonin reuptake inhibitors, tricyclic antidepressants, sildenafil).
* Reported cancer-related fibromyalgia or neuropathic pain conditions
* Have a medical contraindication to, or prior serious adverse events from, cannabis or brownie ingredients (e.g., food sensitivities to gluten/wheat, chocolate, eggs)
* Consume the equivalent of >2 cups of coffee/day (to reduce variability related to metabolic interactions with caffeine)
* Have any of the following: uncontrolled hypertension (i.e., systolic >140 mm Hg and/or diastolic >90 mm Hg on three separate occasions; systolic >170 or diastolic >110 on any occasion), liver function tests >3 times normal, blood urea Nitrogen and Creatinine outside normal range
* Have a physical limitation that will interfere with completing study tasks
* Have child-bearing potential (women)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Vital Signs - Blood Pressure | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  systolic/diastolic blood pressure (mmHg)
Vital Signs - Respiration | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  respiration rate (breaths per minute)
Vital Signs - Pulse | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  pulse (beats per minute)
Self/Observer Ratings - Pain | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  Visual Analog Scales (making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain")
Self/Observer Ratings - Side Effects | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  Side Effects Ratings
Self/Observer Ratings - POMS | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  Profile of Mood States (POMS) short form - using a five-point scale ranging from "not at all" to "extremely."
Self/Observer Ratings - CADSS | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  Clinician Administered Dissociative Symptoms Scale (CADSS)-
Self/Observer Ratings - PROMIS | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  Patient Reported Outcomes Measurements Information System (PROMIS) Cognitive Function short form v2
Balance Tests - Four-Stage | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  The Four-Stage Balance Test- When the patient is steady, let go, and time how long they can maintain the position, but remain ready to assist the patient if they should lose their balance.
Balance Tests - Timed Up and Go | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  The Timed Up & Go Test- Timing commences on the command 'go' and stops when the subject's back is positioned against the back of the chair after sitting down.
Balance Tests - 30 sec chair-stand | pre-drug and 1, 2, 3, and 5.5 hours post-drug administration
  The 30-Second Chair-Stand Test- the number of times the patient comes to a full standing position in 30 seconds.

SECONDARY OUTCOMES:
Cognitive Function Tests - Flanker | pre-drug and 3 hours post-drug administration
  Flanker inhibitory control and attention test- participants are required to indicate the left-right orientation of a centrally presented stimulus while inhibiting attention to the potentially incongruent stimuli that surround it
Cognitive Function Tests - Picture Sequence | pre-drug and 3 hours post-drug administration
  Picture sequence memory- Participants are shown a number of activities, and then asked to reproduce the sequence of pictures as it was presented to them.
Cognitive Function Tests - Sorting | pre-drug and 3 hours post-drug administration
  List sorting working memory -a sequencing task requiring to sort information and sequence it
Cognitive Function Tests - Vocab | pre-drug and 3 hours post-drug administration
  Picture vocabulary test- to measure the receptive (hearing) vocabulary of English-speaking adults
Cognitive Function Tests - Oral Reading | pre-drug and 3 hours post-drug administration
  Oral reading recognition test- participants see a letter or word onscreen and must pronounce or identify it.
Cognitive Function Tests - Card Sort | pre-drug and 3 hours post-drug administration
  Dimensional change card sort test- participants switch from sorting cards one way (e.g., by color) to sorting them a different way (e.g., by shape)
Cognitive Function Tests - pattern processing | pre-drug and 3 hours post-drug administration
  Pattern comparison processing speed test- measures speed of processing by asking participants to discern whether two sideby-side pictures are the same or not.
Cognitive Function Tests - Auditory learning | pre-drug and 3 hours post-drug administration
  Auditory learning verbal test- Five presentations of a 15-word list are given, each followed by attempted recall.
Cognitive Function Tests - Oral symbol | pre-drug and 3 hours post-drug administration
  Oral symbol digit test- given 120 seconds to orally match symbols with digits as quickly as possible.

OTHER OUTCOMES:
Acceptability - session length | 1 day after sessions 1, 2, and 3
  session length- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - ride service | 1 day after sessions 1, 2, and 3
  ride service- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - types of assessments | 1 day after sessions 1, 2, and 3
  types of assessments- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - frequency of assessments | 1 day after sessions 1, 2, and 3
  frequency of assessments- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - duration of assessments | 1 day after sessions 1, 2, and 3
  duration of assessments- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - wait times | 1 day after sessions 1, 2, and 3
  wait times- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability- activities | 1 day after sessions 1, 2, and 3
  activities between assessment cycles- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - food | 1 day after sessions 1, 2, and 3
  food- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])
Acceptability - AEs | 1 day after sessions 1, 2, and 3
  Adverse Events- Likert Scale (0 [not at all acceptable]-5 [completely acceptable])

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No